CLINICAL TRIAL: NCT07150507
Title: Effectiveness of Breathing Therapy in Reducing Sleep and Fatigue Symptoms in Patients With Schizophrenia
Brief Title: The Effectiveness of Breathing Therapy in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mine CENGİZ, Lecturer Physician, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCENGİZ6
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breathing Therapy
Keywords: Breathing Therapy; Schizophrenia patients; Sleep; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Session 1: Preparatory Session (Experimental): *Meeting the patients *Introducing the content of psychoeducation *Emphasizing the importance of regular and timely attendance at training *Determining training dates *Sharing individuals' experiences and expectations
  Interventions: Other: Session 1: Preparation Session
- Session 2: Recognizing the Illness (Experimental): *What is schizophrenia? *What are its symptoms? *What does treatment involve?
  Interventions: Other: Session 2: Recognizing the Illness
- Session 3: Evaluating Treatment (Experimental): *Considerations regarding medication use *Side effects of medication use *Exacerbations in schizophrenia *Premonitory symptoms.
  Interventions: Other: Session 3: Treatment Evaluation
- Session 4: *What is anger? (Experimental): *What are the symptoms of anger? *What are the methods for coping with anger?
  Interventions: Other: Session 4: What is anger?
- Session 5: Communication *What is communication? (Experimental): *The importance of communication. *Fundamentals of communication, self-language practice *Ways to prevent communication difficulties.
  Interventions: Other: Session 5: Communication
- Session 6: What is relaxation? (Experimental): What is progressive relaxation. Relaxation CD introduction
  Interventions: Other: Session 6: What is relaxation?
- Session 7: Relaxation (Experimental): Performing the relaxation CD with patients
  Interventions: Other: Session 7: Relaxation
- Session 8: Evaluation (Experimental): *Reinforcement of what has been learned. *Evaluation of the program. *Receiving feedback
  Interventions: Other: Session 8: Evaluation

INTERVENTIONS:
Other: Session 1: Preparation Session — *Meeting Patients *Introducing the Content of Psychoeducation *Emphasizing the Importance of Regular and Timely Attendance at Training *Determining Training Dates *Sharing Individuals' Experiences and Expectations
  Arms: Session 1: Preparatory Session
Other: Session 2: Recognizing the Illness — *What is Schizophrenia? *What are its Symptoms? *What Does Treatment Include?
  Arms: Session 2: Recognizing the Illness
Other: Session 3: Treatment Evaluation — *Things to Consider When Using Medication *Side Effects of Medication *Exacerbation of Schizophrenia *Precursor Symptoms.
  Arms: Session 3: Evaluating Treatment
Other: Session 4: What is anger? — *What are the symptoms of anger? *What are the methods for coping with anger?
  Arms: Session 4: *What is anger?
Other: Session 5: Communication — *What is communication? *The importance of communication. *Fundamentals of communication, working on "I" language. *Ways to prevent communication difficulties.
  Arms: Session 5: Communication *What is communication?
Other: Session 6: What is relaxation? — What is progressive relaxation? Introducing a relaxation CD
  Arms: Session 6: What is relaxation?
Other: Session 7: Relaxation — Practicing the relaxation CD with patients
  Arms: Session 7: Relaxation
Other: Session 8: Evaluation — *Reinforcing what has been learned. *Evaluating the program. *Obtaining feedback
  Arms: Session 8: Evaluation

SUMMARY:
This study aimed to determine the effects of breathing therapies on sleep disturbances and fatigue in patients with schizophrenia.The study will be conducted at a CMHC in Ağrı province between May and August 2021. At the CMHC, community-based mental health services are provided to patients with severe mental disorders (schizophrenia, bipolar disorder) who are in remission as assessed by a psychiatrist. The study is planned to be conducted with patients who meet the study criteria, without using a sample selection method. Patients over the age of 18 registered with CMHC and followed with a diagnosis of schizophrenia were contacted by phone and invited to CMHC. The study was conducted with patients who met the inclusion criteria and agreed to participate. Data will be collected using the Descriptive Characteristics Form, the DSM-5 Sleep Disorder Scale, and the Brief Fatigue Inventory. The experimental group received eight sessions of respiratory therapy.The control group received no intervention. The study sample size was calculated using the GPower computer program. A power analysis performed at α=0.05 revealed an effect size of 150.153 (d=0.8), providing 90% power. Therefore, it was calculated that a minimum of 68 patients should be included in the sample.

DETAILED DESCRIPTION:
Study data were collected by the researcher through face-to-face interviews. The study included individuals diagnosed with schizophrenia who met the inclusion criteria (registration in a CMHC, having a diagnosis of schizophrenia, willingness to participate in the study, and openness to communication and collaboration). Pre-test measurement instruments were administered to the participants. The experimental group received eight sessions of respiratory therapy. The control group received no intervention. Post-test data were collected following the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with a CMHC
* Being diagnosed with schizophrenia
* Being between the ages of 18 and 60
* Being willing to participate in the study
* Being open to communication and cooperation
* Being in remission

Exclusion Criteria:

* Not being open to communication and cooperation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | up to 1 day
  It consists of a total of 8 questions (age, gender, marital status, education level, duration of illness, income status, family history of mental illness and employment status) created by the researcher in the light of literature and includes the sociodemographic characteristics of the patients.

SECONDARY OUTCOMES:
DSM-5 Sleep Disorder Scale | up to 1 day
  The DSM-5 Sleep Disorder Adult Scale Short Form is an eight-item scale that assesses sleep disturbances in individuals aged 18 and older. The scale is designed to be completed by the individual before a clinician's consultation. Each item asks the patient (or an informed person) to rate the severity of their sleep disturbance over the past seven days. The scale's validity and reliability in Turkish were conducted by Yüzeren et al. in 2017.

OTHER OUTCOMES:
Brief Fatigue Inventory | up to 1 day
  Developed by Mendoza and colleagues at the M.D. Anderson Cancer Center in 1999, the scale consists of 10 questions. The form assesses general fatigue levels (fatigue felt at the time of the interview, general fatigue experienced within the last 24 hours, and the worst fatigue level experienced within the last 24 hours) and the degree to which daily activities (general activity, mood, walking ability, life outside the home, communication with others, and joy of life) have been affected by fatigue in the last 24 hours. The arithmetic mean of the scores given for these first three questions is calculated to obtain each individual's fatigue score. The Cronbach's α value for the original scale, developed by Mendoza and colleagues (1999), was found to be 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Cengiz lecturer doctor, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided